CLINICAL TRIAL: NCT03900494
Title: Comparing the Efficacy of Two Valved Holding Chambers for Bronchodilator Administration in 0.5-4 Years Old Children With Acute Wheezing - a Randomized Clinical Trial
Brief Title: Comparing the Efficacy of Two Valved Holding Chambers in Acute Wheezing
Acronym: CHAMBER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Kuopio University Hospital (Other); Oulu University Hospital (Other); Tampere University Hospital (Other); Terveystalo Healthcare Services (Unknown)
Responsible Party: Principal Investigator, Peter Csonka, Specialist in pediatrics and pediatric allergology, Tampere University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ETL-R19030
Record Dates: First submitted 2019-03-29; First posted 2019-04-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Bronchitis Obstructive; Bronchiolitis; Obstruction; Bronchospasm; Bronchitis
Keywords: salbutamol; valved holding chamber; pMDI; inhalation therapy; children; toddlers; emergency room; bronchitis; bronchiolitis
MeSH Terms: conditions — Bronchiolitis; Bites and Stings; Bronchial Spasm; Bronchitis; Emergencies

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children treated with VHC 1 (Active Comparator): In this group children are receiving salbutamol with valved holding chamber number 1. Otherwise the children in both groups are treated exactly the same way. The only difference is the device used to deliver the bronchodilator. Children in both arms have the same condition and the same inclusion and exclusion criteria. We only compare the efficacy of the two VHC devices.
  Interventions: Device: VHC 1
- Children treated with VHC 2 (Active Comparator): In this group children are receiving salbutamol with valved holding chamber number 2. Otherwise the children in both groups are treated exactly the same way. The only difference is the device used to deliver the bronchodilator. Children in both arms have the same condition and the same inclusion and exclusion criteria. In this group children are receiving salbutamol with valved holding chamber number 1. Otherwise the children in both groups are treated exactly the same way. The only difference is the device used to deliver the bronchodilator. Children in both arms have the same condition and the same inclusion and exclusion criteria.
  Interventions: Device: VHC 2

INTERVENTIONS:
Device: VHC 1 — Salbutamol 0.6-0.8 mg given 20-40 min. maximum four times depending on the bronchodilator response delivered via valved holding chamber 1. Same salbutamol dosing protocol for both arms. Only difference is the VHC used.
  Arms: Children treated with VHC 1
Device: VHC 2 — Salbutamol 0.6-0.8 mg given 20-40 min. maximum four times depending on the bronchodilator response delivered via valved holding chamber 2. Same salbutamol dosing protocol for both arms. Only difference is the VHC used.
  Arms: Children treated with VHC 2

SUMMARY:
The incidence of physician confirmed asthma is approximately 4-7% in children. An additional 5% of children suffer from infection-related bronchiolitis and obstructive bronchitis. Of all patient visits at pediatric emergency rooms, 1 out of 10 is due to breathing difficulties with a great proportion leading to hospitalization.

Salbutamol is the most commonly used drug in the treatment in acute bronchial obstruction. A vast majority of children require a spacer device (valved holding chamber, VHC) for the delivery of the drug aerosol. There are several different types of VHC on the market, but no recommendations on the device selection have been published. Both in in vivo and in vitro studies significant differences between different spacer devices have been reported.

The study compares two different VHCs in the treatment of acute breathing difficulties in children. The end-points in this randomized physician-blinded study are symptom relief, rate of hospitalization, symptom recurrence, treatment compliance, and adverse events.

The study will be conducted in pediatric emergency rooms (ER) in three university hospitals in Finland and one private clinic that routinely treat this type of patients. The treatment is given according to national treatment guidelines and no blood samples are drawn for study purposes. Both of the VHCs used in this study have been approved for use in clinical practice.

DETAILED DESCRIPTION:
This study compares two valved holding chamber (VHC) devices in the treatment of acute airway obstruction in children. Eighty children (6 months to 4 years of age) will be recruited with moderate to severe dyspnea according to the Respiratory Distress Assessment Instrument (RDAI score ≥6). After receiving an informed consent from the parents/caregivers, the child is randomized to receive treatment with either Babyhaler® or Optichamber Diamond® VHC. Patients with underlying medical conditions listed in the study protocol, patients requiring immediate hospitalization or not willing to participate will be excluded from the study. Information on the medical history together with treatment response will be recorded using a manual case report form. According to calculations of the statistical power using the RDAI-score as an end-point, a total of 80 patients (40 patients in both study groups) are needed for the study.

The study hypothesis is that the two VHCs are not equally efficient in treating acute shortage of breath in children aged 0.5-4 years.

ELIGIBILITY:
Inclusion Criteria:

- Children (age 0.5-4 years) seeking medical aid due to respiratory distress caused by bronchial obstruction

Exclusion Criteria:

* requiring immediate admission to inpatient treatment in hospital
* peripheral capillary oxygen saturation below 85% on admission
* physician-confirmed pneumonia
* inspiratory crackles on lung auscultation
* croup
* airway foreign body
* impaired renal or liver function
* immune compromised patient
* general condition affecting the study per investigation judgement
* bronchopulmonary dysplasia
* long-acting beta-adrenoceptor agonist treatment
* recruited to the ongoing study earlier
* have been enrolled in a clinical trial within 30 days prior to admission
* not willing to participate

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Number of subjects whose RDAI symptom score decrased by 2 or more | 20 minutes after the second salbutamol-dose and if necessary 20 minutes after the third or fourth salbutamol-dose. Maximum 5 hours.
  Respiratory Distress Assessment Instrument (RDAI) score. Change from baseline at each evaluation point. Discharge time is dependent on the score at each evaluation point. Minimum score 0 (best), maximum score 17 (worst). Inclusion criteria is at least 6.
Difference in the mean capillary oxygen saturation change between groups | 20 minutes after the second salbutamol-dose and if necessary 20 minutes after the third or fourth salbutamol-dose. Maximum 5 hours.
  Peripheral capillary oxygen saturation (%). Change from baseline at each evaluation point. Minimum 85 % (if below, not suitable for the study), maximum 100 %.
Difference in the mean respiratory rate change between group | 20 minutes after the second salbutamol-dose and if necessary 20 minutes after the third or fourth salbutamol-dose. Maximum 5 hours.
  Respiratory rate per minute. Change from baseline at each evaluation point. Minimum N/A, maximum N/A.

SECONDARY OUTCOMES:
Compliance to treatment, compared between groups | Throughout the ER visit. Maximum 5 hours.
  Compliance to the treatment using a structured questionnaire conducted both by the parents and by the nurses treating the child in the emergency room.
  Cooperation score from 0 to 5: 0 = no measurement possible; 1 = continuously crying, screaming, or struggling against the procedure; 2 = crying, screaming, or struggling, but not continuously; 3 = not very good cooperation, but no crying or screaming; 4 = good cooperation, but clearly not comfortable; 5 = good cooperation and quiet breathing during the whole measurement.
Number of subjects hospitalized in both group | After the last dose of salbutamol. Maximum 5 hours.
  The information on whether the patient is discharged from the emergency room or admitted to hospital for further treatment will be recorded in the case report form.
Number of drug doses given in both groups | Throughout the ER visit. Maximum 5 hours.
  Number of salbutamol-doses given to the patient. Minimum two, maximum four doses. Less dose is better.
Difference in the mean heart rate change between groups | After each salbutamol dose. Maximum 5 hours.
  Change in heart rate per minute. Minimum N/A, maximum N/A.

CONTACTS AND LOCATIONS:
Locations (4):
- Finland (4):
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Terveystalo Tampere, Tampere
  - Tampere University Hospital, Tampere

IPD SHARING:
Plan to Share IPD: Undecided